CLINICAL TRIAL: NCT00852033
Title: Alcohol Early Intervention for Freshmen
Acronym: Transitions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Mark D. Wood, University of Rhode Island
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: NIAAA-Wood-AA013919; NIH Grant 5R01AA013919-04
Record Dates: First submitted 2009-02-24; First posted 2009-02-26 (Estimated); Last update posted 2009-02-26 (Estimated); Status verified 2009-02

CONDITIONS: Alcohol Abuse
Keywords: alcoholism; alcohol abuse; prevention; behavior modification; parent offspring interaction; university student; substance abuse related behavior; adolescence
MeSH Terms: conditions — Alcoholism | interventions — Immunization, Secondary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (No Intervention): Assessment Group (no intervention)
  Interventions: Other: Assessment only
- 2 (Active Comparator): Brief Motivational Intervention (BMI)
  Interventions: Behavioral: Brief Motivational Intervention (BMI)
- 3 (Active Comparator): Parent Based Intervention (PBI)
  Interventions: Behavioral: Parent Based Intervention plus booster
- 4 (Active Comparator): BMI and TBI
  Interventions: Behavioral: Brief Motivational Intervention (BMI); Behavioral: Parent Based Intervention plus booster; Behavioral: Combined brief motivational intervention and parent based intervention plus boosters for both interventions

INTERVENTIONS:
Behavioral: Brief Motivational Intervention (BMI) — Students met with trained interventionists. The initial BMI took place during the fall semester of the freshmen year for approximately 45 minutes. Individualized feedback was used to guide the BMI sessions. The feedback data were gathered through an online survey completed within two weeks of the scheduled appointment to ensure the use of proximal feedback reflecting current drinking. Feedback was tailored so that drinkers received information on their personal drinking patterns, heavy episodic drinking, and alcohol-related consequences, and abstainers received feedback on their perceived barriers for maintaining abstinence, the safety and health benefits of their choice not to drink, and their experience with second-hand effects of alcohol use. In the spring of the freshmen year, students received a BMI 'booster' session. Individualized feedback was created from the original online survey and the 10 month follow-up assessment.
  Other Names: BMI
  Arms: 2; 4
Behavioral: Parent Based Intervention plus booster — The PBI is a handbook-based intervention modified from Turrisi and colleagues (2001). It was designed to raise parental awareness of alcohol abuse and consequences among college students and increase parental effort to address this issue with their teen.
  Other Names: PBI
  Arms: 3; 4
Behavioral: Combined brief motivational intervention and parent based intervention plus boosters for both interventions — A combination of Intervention 1 and 2.
  Arms: 4
Other: Assessment only — No intervention, assessment only.
  Arms: 1

SUMMARY:
Alcohol abuse among college students is a significant and long-standing public health issue. The transition into college is marked by substantial increases in alcohol abuse and problems, suggesting the importance of interventions that take place prior to and immediately following matriculation. To date, early interventions with this population have yielded modest results with very little evidence identifying either the factors that are responsible for observed effects or specific individual or situational factors that qualify intervention efficacy. There is preliminary evidence for the efficacy of individualized feedback (IF) in reducing college student alcohol abuse. Additionally, a sizeable body of research with early adolescents and emerging work with college students point to the utility of parent-based interventions (PBI). The major aim of this research is to provide the first test of the unique and combined efficacy of these two successful interventions in reducing alcohol abuse among matriculating college students.

DETAILED DESCRIPTION:
Using a 2 X 2 IF (yes; no) X PBI (yes; no) factorial design, this study will determine whether IF and PBI with "boosters" are effective in reducing alcohol abuse among incoming college students. It is hypothesized that groups receiving IF and PBI will demonstrate lower levels of alcohol abuse over the first two years of college than those not receiving these interventions and that the effects of combining these interventions will be additive (Specific Aim 1). Structural equation modeling techniques will be used to conduct mediational analyses investigating theoretically derived hypotheses about the processes by which intervention factors influence alcohol use and problems (Specific Aim 2). Hierarchical multiple regression analyses will examine hypothesized individual and situational moderators of intervention efficacy (Specific Aim 3). The use of a factorial design and explicit mediational analyses will allow for very strong inferences regarding the "active ingredients" of intervention efficacy. The long-term objectives of this research are to improve the efficacy of early interventions and to inform research and theory on the etiology of alcoholism. More effective interventions, particularly those that target students during a developmental transition of enhanced risk, will result in fewer injuries from acute intoxication, enhance retention and learning, and lessen the development of alcoholism as a result of chronic alcohol abuse.

ELIGIBILITY:
Inclusion Criteria:

* All incoming students who paid their university attendance deposit by May 1st of the recruitment years were eligible for participation.

Exclusion Criteria:

* transfer students,
* married,
* not living with a parent/guardian,
* returning students older than 20 years
* reached the alcohol use cut-off criteria (40 or more drinks per week and two symptoms of alcohol dependence)

Ages: 17 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1014 (Actual)
Dates: Start 2004-01; Primary Completion 2007-06 (Actual); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
Daily Drinking Questionnaire | Baseline, 10 months, 22months, 46 months
Young Adult Problems Screening Test "YAAPST" | Baseline, 10 months, 22months, 46months

CONTACTS AND LOCATIONS:
Overall Officials: Mark D Wood, PhD, Principal Investigator — University of Rhode Island
Locations (1):
- University of Rhode Island, Department of Psychology, Kingston, Rhode Island, United States